CLINICAL TRIAL: NCT01630486
Title: KoreaN Cohort Study for Outcome in Patients With Chronic Kidney Disease
Brief Title: KoreaN Cohort Study for Outcome in Patients With Chronic Kidney Disease : A 10-year Longitudinal Cohort Study of the Chronic Kidney Disease
Acronym: KNOW-CKD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kook-Hwan Oh, Professor, Seoul National University Hospital
Other Study IDs: KNOW-CKD
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Disease
Keywords: renal progression; mortality; complications; risk factors; role of biochemical parameters; genetic influence
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A biobank is also established for the DNA, serum and urine taken at regular interval.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- glomerulonephritis: adult CKD patients, whose underlying etiology is glomerulonephritis, either clinically diagnosed or pathologically proven
- hypertensive nephropathy: adult CKD patients, whose underlying etiology is hypertensive nephropathy
- polycystic kidney disease: adult CKD patients, whose underlying etiology is autosomal dominant polycystic kidney disease
- diabetic nephropathy: adult CKD patients, whose underlying etiology is diabetic nephropathy

SUMMARY:
The goals of the KNOW-CKD (KoreaN cohort study for Outcome in patients With Chronic Kidney Disease) study are 1) to establish a CKD cohort representing Korean CKD population for up to 10-year follow-up, and 2) to investigate the renal progression, mortality, complications, risk factors, role of biochemical parameters and the genetic influence.

KNOW-CKD Research Group comprises nephrologists, pediatric nephrologists, epidemiologists and statisticians from eleven centers in Korea. KNOW-CKD will enroll 2,850 individuals with CKD stage from 1 to 5 between 2011 and 2015 and follow them up to 10 years. Dialyzed patients or those with allograft kidney are excluded. At enrollment and at pre-specified intervals, laboratory tests will be conducted on the kidney function, biochemical profiles, anemia, cardiovascular complication (echocardiography, coronary CT, arterial stiffness), and mineral bone disorder. A biobank is also established for the DNA, serum and urine at regular interval. Information on the medical history, health questionnaires, QoL will also be collected. Web-based case-report forms (CRF) is developed for the systemic management of the patient data.

ELIGIBILITY:
Inclusion Criteria:

* Age: >20 and <75 yr,
* CKD stage 1 through 5
* predialysis

Exclusion Criteria:

* Unable or unwilling to give consent
* Previously received chronic dialysis
* Previous any organ transplant
* Heart failure
* Known liver cirrhosis
* past or current cancer
* Pregnant women
* Single kidney due to trauma or donation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD stage 1 through 5 Ages below 75
Sampling Method: Non-Probability Sample
Enrollment: 2238 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
overall mortality | 10 years

SECONDARY OUTCOMES:
cardiovascular event | 10 years
renal replacement therapy | 10 years
  dialysis or kidney transplantation
doubling of serum creatinine | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park CH, Kim HW, Park JT, Chang TI, Yoo TH, Oh KH, Anderson AH, Yang W, Cohen JB, Rahman M, Kang SW, Han SH; on the behalf of CRIC Study and KNOW-CKD Investigators. BP and Kidney Disease Progression in Advanced CKD: Findings from the Chronic Renal Insufficiency Cohort and KoreaN Cohort Study for Outcome in Patients with CKD Studies. Clin J Am Soc Nephrol. 2025 Jun 6;20(9):1179-1189. doi: 10.2215/CJN.0000000760. PMID 40478754
- [Derived] Park CH, Kim HW, Joo YS, Park JT, Chang TI, Yoo TH, Park SK, Chae DW, Chung W, Kim YS, Oh KH, Kang SW, Han SH; on the behalf of the KNOW-CKD (Korean Cohort Study for Outcomes in Patients With Chronic Kidney Disease) Investigators. Association Between Systolic Blood Pressure Variability and Major Adverse Cardiovascular Events in Korean Patients With Chronic Kidney Disease: Findings From KNOW-CKD. J Am Heart Assoc. 2022 Jun 7;11(11):e025513. doi: 10.1161/JAHA.122.025513. Epub 2022 Jun 3. PMID 35656977
- [Derived] Kim JY, Park JT, Kim HW, Chang TI, Kang EW, Ahn C, Oh KH, Lee J, Chung W, Kim YS, Kim SW, Yoo TH, Kang SW, Han SH; KNOW-CKD (Korean Cohort Study for Outcomes in Patients With Chronic Kidney Disease) Investigators. Inflammation Alters Relationship Between High-Density Lipoprotein Cholesterol and Cardiovascular Risk in Patients With Chronic Kidney Disease: Results From KNOW-CKD. J Am Heart Assoc. 2021 Aug 17;10(16):e021731. doi: 10.1161/JAHA.120.021731. Epub 2021 Aug 7. PMID 34369187
- [Derived] Lee C, Park KH, Joo YS, Nam KH, Chang TI, Kang EW, Lee J, Oh YK, Jung JY, Ahn C, Lee KB, Park JT, Yoo TH, Kang SW, Han SH. Low High-Sensitivity C-Reactive Protein Level in Korean Patients With Chronic Kidney Disease and Its Predictive Significance for Cardiovascular Events, Mortality, and Adverse Kidney Outcomes: Results From KNOW-CKD. J Am Heart Assoc. 2020 Nov 3;9(21):e017980. doi: 10.1161/JAHA.120.017980. Epub 2020 Oct 23. PMID 33092438
- [Derived] Kim HJ, Lee J, Chae DW, Lee KB, Sung SA, Yoo TH, Han SH, Ahn C, Oh KH. Serum klotho is inversely associated with metabolic syndrome in chronic kidney disease: results from the KNOW-CKD study. BMC Nephrol. 2019 Apr 3;20(1):119. doi: 10.1186/s12882-019-1297-y. PMID 30943913
- [Derived] Chae SY, Chung W, Kim YH, Oh YK, Lee J, Choi KH, Ahn C, Kim YS. The Correlation of Serum Osteoprotegerin with Non-Traditional Cardiovascular Risk Factors and Arterial Stiffness in Patients with Pre-Dialysis Chronic Kidney Disease: Results from the KNOW-CKD Study. J Korean Med Sci. 2018 Dec 11;33(53):e322. doi: 10.3346/jkms.2018.33.e322. eCollection 2018 Dec 31. PMID 30595681
- [Derived] Kang E, Lee J, Kim HJ, Han M, Kim SW, Lee KB, Sung S, Yoo TH, Chung W, Ahn C, Oh KH. The association between socioeconomic disparities and left ventricular hypertrophy in chronic kidney disease: results from the KoreaN Cohort Study for Outcomes in Patients With Chronic Kidney Disease (KNOW-CKD). BMC Nephrol. 2018 Aug 16;19(1):203. doi: 10.1186/s12882-018-1005-3. PMID 30115015
- [Derived] Kim HJ, Kang E, Oh YK, Kim YH, Han SH, Yoo TH, Chae DW, Lee J, Ahn C, Oh KH. The association between soluble klotho and cardiovascular parameters in chronic kidney disease: results from the KNOW-CKD study. BMC Nephrol. 2018 Mar 5;19(1):51. doi: 10.1186/s12882-018-0851-3. PMID 29506503
- [Derived] Lee MJ, Park JT, Park KS, Kwon YE, Han SH, Kang SW, Choi KH, Oh KH, Park SK, Chae DW, Lee K, Hwang YH, Kim SW, Kim YH, Kang SW, Lee J, Ahn C, Yoo TH. Normal body mass index with central obesity has increased risk of coronary artery calcification in Korean patients with chronic kidney disease. Kidney Int. 2016 Dec;90(6):1368-1376. doi: 10.1016/j.kint.2016.09.011. PMID 27884313
- [Derived] Han JS, Lee MJ, Park KS, Han SH, Yoo TH, Oh KH, Park SK, Lee J, Hyun YY, Chung W, Kim YH, Ahn C, Choi KH. Albuminuria as a Risk Factor for Anemia in Chronic Kidney Disease: Result from the KoreaN Cohort Study for Outcomes in Patients With Chronic Kidney Disease (KNOW-CKD). PLoS One. 2015 Oct 2;10(10):e0139747. doi: 10.1371/journal.pone.0139747. eCollection 2015. PMID 26430892
- [Derived] Oh KH, Park SK, Park HC, Chin HJ, Chae DW, Choi KH, Han SH, Yoo TH, Lee K, Kim YS, Chung W, Hwang YH, Kim SW, Kim YH, Kang SW, Park BJ, Lee J, Ahn C; Representing KNOW-CKD Study Group. KNOW-CKD (KoreaN cohort study for Outcome in patients With Chronic Kidney Disease): design and methods. BMC Nephrol. 2014 May 19;15:80. doi: 10.1186/1471-2369-15-80. PMID 24884708